CLINICAL TRIAL: NCT06157671
Title: The LINFU® (A Noninvasive Method for Increasing Exfoliation of Pancreatic Ductal Cells Into Pancreatic Fluid) U.S. Registry for the Detection of Low and High- Grade Atypia and Early, Asymptomatic Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: The LINFU® U.S. Registry for the Detection of Asymptomatic Pancreatic Ductal Adenocarcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Adenocyte, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Adenocyte 101
Record Dates: First submitted 2023-11-12; First posted 2023-12-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Intraepithelial Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Slides and cell blocks made from pancreatic fluid collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients at increased risk for developing pancreatic cancer: Patients being screened for pancreatic cancer because they have known risk factors (i.e. smoking, diabetes, chronic pancreatitis, family history of pancreatic cancer, or certain genetic syndromes) and are undergoing other imaging diagnostic tests to determine if they have pancreatic cancer

SUMMARY:
Adenocyte has developed LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) as a method of identifying early, asymptomatic pancreatic cancer and its noninvasive precancerous lesions. The test involves ultrasound and an analysis of pancreatic juice. A neural network-based computer-assisted system may be utilized to enhance the analysis. Patients enrolled are being screened for pancreatic cancer because they have known risk factors (i.e. smoking, diabetes, chronic pancreatitis, family history of pancreatic cancer, or certain genetic syndromes).

DETAILED DESCRIPTION:
Adenocyte has developed a proprietary pancreatic cancer detection method, LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) to increase the sensitivity of pancreatic juice cytology. LINFU® consists of analysis of pancreatic fluid collected with the help of low intensity non-focused ultrasound excitation of the pancreas. A contrast agent will be used to create bubbles and possibly increase the number of pancreatic cell we collect for the study. Secretin is also used to increase the number of pancreatic cell excretion to maximize the number of cells collected. A neural network-based computer-assisted system may be used to enhance the analysis of specimens.

In this registry, LINFU® will be studied in patients who are at increased risk for developing pancreatic cancer including those being screened because they have known risk factors (i.e. smoking, diabetes, chronic pancreatitis, family history of pancreatic cancer, or certain genetic syndromes) and are undergoing other diagnostic tests (i.e. EUS- FNA, MRI/MRCP, ERCP, CT, CEUS).

In this registry, a standardized Case Report Form will be completed for every subject enrolled. Information obtained at baseline will include patient history, clinical and demographic information including relevant comorbidities and pancreatic disease history, and screening and pathology test results. The results of all diagnostic tests, surgeries, and biopsies performed after the LINFU® technique for a period of 5 years will be recorded and maintained as clinical registry data. This includes testing and procedures received since enrollment including EUS- FNA, MRI/MRCP, ERCP, CT, CEUS, treatments performed, pathology results, and pancreatic disease history since enrollment.

The registry case report form is the primary data collection instrument for the registry. All data requested on the form must be recorded and these forms will be monitored carefully by the sponsor to ensure they are completely filled out properly.

.

ELIGIBILITY:
Inclusion Criteria

* Both males and females will be enrolled and must be at least 18 years of age under age of 90
* Patients who, in the opinion of the Investigator, are at elevated risk of developing a pancreatic malignancy because they have known risk factors for PDAC.
* High risk asymptomatic patients being screened for PDAC.
* All patients must undergo contemporaneous imaging (within 90 days of LINFU®) with one or more of the following: EUS± FNA, MRI/MRCP, ERCP, CT or CEUS.
* Institutional Review Board (IRB)-approved consent must be signed by patients to participate in this study.

Exclusion Criteria:

* Patient under the age of 18 and over the age 90
* Contraindications to LINFU®/EUS/ERCP as determined by study investigators including: patient with uncorrectable coagulopathy; patient that cannot undergo anesthesia due to cardiopulmonary contraindication as deemed by the anesthesiologist; unstable medically (cardiopulmonary, neurologic, or cardiovascular status)
* Patients with clinical signs or symptoms of PDAC
* Patients undergoing EUS or ERCP for a suspected bile duct cancer arising from the intrahepatic or extrahepatic biliary epithelium
* Patients with documented intraductal papillary mucinous neoplasm of the pancreas (IPMN)
* Pregnant females will be excluded
* Patient that is unable to provide informed consent
* Patient with known allergy to the microbubble contrast agent or secretin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk asymptomatic patients being screened for pancreatic cancer who are scheduled for EUS± FNA, MRI/MRCP, ERCP, CT or CEUS will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® will be compared to standard screening methods | 5 years
  The total number of asymptomatic pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® by analysis of pancreatic fluid will be compared to the number of these lesions identified with current screening tests, including EUS- FNA, MRI/MRCP, ERCP, CT and CEUS.

SECONDARY OUTCOMES:
The change in size of pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® will be determined over a 5 year period. | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS to assess whether these tumors increase in size (measured in mm) and to determine how many require medical or surgical intervention.
Determine the number of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® that require medical or surgical intervention. | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS to assess whether these tumors increase how many require medical or surgical intervention.

OTHER OUTCOMES:
Yearly survival rate of patients with early pancreatic ductal adenocarcinomas or their noninvasive precursor lesions identified only with LINFU® | 5 years
  Patients will be followed by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS and yearly survival rates of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, MD FRCP, Principal Investigator — Manhattan Endoscopy Center
Locations (1):
- Manhattan Endoscopy Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No